CLINICAL TRIAL: NCT01592435
Title: Carestream Digital Radiography Long Length Imaging Manual Stitch Editor Software Data Collection
Brief Title: Carestream Digital Radiography Long Length Imaging Software Data Collection Protocol
Acronym: LLI-MSE
Status: Completed | Type: Observational
Sponsor: Carestream Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 8H9323
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Spinal Injuries
MeSH Terms: conditions — Spinal Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pred. & Invest.-All Study Participants: Cedera AccuStitch Software is standard of care software currently used at sites.
  Carestream DR LLI software is investigational software used for reconstruction.

SUMMARY:
The study objective is to acquire composite images generated by the Carestream Long Length Imaging (LLI) software and demonstrate that the images stitched using the Carestream LLI software and the images stitched using a approved predicate device are acceptable for clinical use.

DETAILED DESCRIPTION:
The study consists of subject enrollment to collect images in a clinical setting, followed by a review of the stitched images by radiologists or qualified orthopedic surgeons to assess overall usability of the composite images.

This study includes clinical data collection of individual (raw and processed) and composite DR images from a Carestream device using alpha rotation to acquire the images. There is no subject involvement other than obtaining informed consent in order to use patient images and Case Record Forms (CRF), including supporting radiology reports. This study has no effect on clinical treatment and no foreseen risks to enrolled subjects.

The predicate software is currently in place at the sites. Carestream will harvest that data and reconstruct with investigational software offsite. A comparison reader study will be performed upon completion of data collection.

Please note this study is considered to be observational because there were no imaging of subject using investigational device. Subjects requiring standard of care diagnostic images were exposed using the commercially available Cedara system. The images captured on the Cedara system were then re-processed using the Carestream investigational software. Subjects gave informed consent for Carestream to reprocess their image data. They did not require any additional imaging using the investigational device.

ELIGIBILITY:
Inclusion Criteria:

* subject has provided informed consent
* Male or Female who require Long Length Imaging

Exclusion Criteria:

* Not able or willing to provide Informed Consent, or consent is withdrawn
* Not able to collect all required case information
* Patients who are unable to stand
* Images which are not clinically acceptable to the user
* Images without a reference object such as a ruler in the image.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects requiring standard of care diagnostic images were exposed using the commercially available Cedara system. The images captured on the Cedara system were then re-processed using the Carestream investigational software. Subjects gave informed consent for Carestream to reprocess their image data. They did not require any additional imaging using the investigational device.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Kirshner, BSRT, Principal Investigator — Heartland Regional Medical Center
Locations (2):
- United States (2):
  - Memorial Medical Center, Springfield, Illinois
  - Heartland Regional Medical Center, Saint Joseph, Missouri

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pred. & Invest.-All Study Participants
Started | 76
Completed | 76
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 76 subjects participated from both sites. 76 image sets were reconstructed with Cedara Accustitch software and the same 76 image sets were reconstructed with Carestream DR LLI software.
Arm/Group | Pred. & Invest.-All Study Participants
Number analyzed (Participants) | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19
  Between 18 and 65 years | 57
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 32

OUTCOME MEASURES:

1. Primary Outcome: Radlex Scale for Diagnostic Capability Ratings - Cedara Accustitch Software (Predicate)
Description: 1-Non-diagnostic - Unacceptable for diagnostic purposes. 2-Limited - Acceptable, with some technical defect. 3-Diagnostic - Image quality that would be expected routinely when imaging cooperative patients. 4-Exemplary - Good, most adequate for diagnostic purposes.
Time Frame: 5 weeks after completion of data collection
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Predicate - Cedera AccuStitch Software: Cedera AccuStitch Software is standard of care software currently used at sites.
Arm/Group | Predicate - Cedera AccuStitch Software
Number analyzed (Participants) | 76
units on a scale | 3.01 (0.04)
Statistical Analysis 1: Comparison: Predicate - Cedera AccuStitch Software; Test type: Superiority or Other; p = 0.02, t-test, 1 sided — level of significance (alpha) = 0.05 All p-values were calculated (and verified) by our statistician and are correct. They were rounded to fit four digits

2. Primary Outcome: Radlex Scale for Diagnostic Capability Ratings - Carestream DR LLI Software (Investigational)
Description: as for outcome 1
Time Frame: 5 weeks after completion of data collection
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Invest. - Carestream DR LLI Software: Carestream DR LLI software is investigational software used for reconstruction.
Arm/Group | Invest. - Carestream DR LLI Software
Number analyzed (Participants) | 76
units on a scale | 3.16 (0.07)
Statistical Analysis 1: Comparison: Invest. - Carestream DR LLI Software; Test type: Superiority or Other; p = 0.00, t-test, 1 sided — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Predicate - Cedera AccuStitch Software: Cedara Accustitch is the standard of care software currently used by sites.
Arm/Group | Predicate - Cedera AccuStitch Software | Invest. - Carestream DR LLI Software
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/76
Other Adverse Events (participants affected / at risk) | 0/76 | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No